CLINICAL TRIAL: NCT04742335
Title: Assessment of Pain, Occupational Fatigue, Sleep and Quality of Life in Nurses
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Doctor Lecturer, Ufuk University
Other Study IDs: 2020-3-17
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Pain in A Joint, Multiple Sites
MeSH Terms: conditions — Arthralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey will be applied to the participants.

SUMMARY:
The aim of the study is to evaluate the pain, occupational fatigue, sleep and quality of life in nurses and the relationships between them. 102 participants working as nurses were included in the study. Data on age, gender, height, weight, working year in the profession, weekly working hours, hand dominance, diagnosed diseases and marital status of the participants were collected. Subsequently, the questions included in the Nordic musculoskeletal questionnaire, occupational fatigue / burnout / recovery scale (OFER), sleep hygiene index (SHI) and World Health Organization quality of life scale (WHOQOL-BREF) questionnaires were answered by the participants.

DETAILED DESCRIPTION:
Nordic Musculoskeletal Questionnaire: It is a scale that evaluates whether symptoms of pain, pain and discomfort have been experienced in the neck, shoulder, elbow, hand-wrist, waist, back, hip-thigh, knee-foot-ankle regions during the last 12 months and whether ordinary indoor and outdoor activities are hampered by these symptoms and whether there has been pain in the mentioned body areas for the last 7 days. It consists of 27 items and each item is answered as yes / no.

Occupational Fatigue Exhaustion Recovery Scale: It is a scale developed to measure occupational fatigue. It consists of 15 items in total and 3 sub-dimensions evaluating chronic fatigue (questions 1-5), acute fatigue (questions 6-10) and recovery (questions 11-15). Each item is scored between 0-6 points (0 = Strongly Disagree, 1 = Disagree, 2 = Somewhat Disagree, 3 = Neither agree nor disagree, 4 = slightly agree, 5 = Agree, 6 = Strongly Agree) by the participants. High scores in the chronic and acute fatigue sub-dimensions mean higher occupational fatigue, and higher scores in the recovery sub-dimension mean better recovery between working periods.

Sleep Hygiene Index: It is a scale that evaluates sleep hygiene. The frequencies of sleep hygiene-related behaviors are questioned in a total of 13 items with a Likert-type scale where each item is scored between 0 and 4 (0 = never, 1 = rarely, 3 = sometimes, 4 = often, 5 = always). Higher scores indicate worse sleep hygiene.

WHOQOL-BREF-TR: It is a scale that evaluates the well-being of individuals in 4 sub-areas in which physical health, psychological status, social relations and environmental conditions are questioned, and their general quality of life and health status with one question. Each item is scored on a 1-5 Likert-type scale. Sub-domain scores represent the quality of life in their field independently of each other. Higher scores indicate better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Working as a nurse

Exclusion Criteria:

* Being under the age of 18
* Having a history of serious trauma and orthopedic surgery in the last 1 year
* Having a chronic severe internal and neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 102 volunteer nurses over 18 years old.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Nordic Musculoskeletal Questionnaire scores | 1 month
  whether symptoms of pain, pain and discomfort have been experienced in the neck, shoulder, elbow, hand-wrist, waist, back, hip-thigh, knee-foot-ankle regions during the last 12 months and whether ordinary indoor and outdoor activities are hampered by these symptoms and whether there has been pain in the mentioned body areas for the last 7 days.
Occupational Fatigue Exhaustion Recovery Scale scores | 1 month
  İt evaluates chronic fatigue, acute fatigue and recovery.
Sleep Hygiene Index score | 1 month
  It evaluates sleep hygiene.
WHOQOL-BREF-TR scores | 1 month
  It evaluates the well-being of individuals in physical health, psychological status, social relations and environmental conditions and their general quality of life and health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)